CLINICAL TRIAL: NCT04938713
Title: Comparison of Ketamine and Esketamine in Ambulatory Patients Treated for Fibromyalgia Syndrome in Pain Clinic. A Single-center, Prospective, Randomized, Double-blind, Crossover Study.
Brief Title: Comparison of Ketamine and Esketamine in Patients Suffering From Fibromyalgia Syndrome.
Acronym: KESK-FIQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Charleroi (Other)
Collaborators: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Brice Constant, MD, MD, Centre Hospitalier Universitaire de Charleroi
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KESK-FIQ
Record Dates: First submitted 2021-06-17; First posted 2021-06-24 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Ketamine; Esketamine; Fibromyalgia Impact Questionnaire; Side effects; Chronic pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Ketamine; Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AB group (Active Comparator): If A = Ketamine and B = Esketamine, each patient included in the study will be randomized in a sequence of administration of the two products. The AB sequence consists of patients starting with intravenous Ketamine 0,3 mg/kg in 1 hour (2 infusions separated by 6 weeks; Period 1) and continuing with intravenous Esketamine 0,15 mg/kg in 1 hour (2 infusions separated by 6 weeks; Period 2). Each patient will be monitored during the IV perfusion, and then, the next hour.
  The patient will receive a total of two infusions of Ketamine and two infusions of Esketamine. Each patient will be his own witness because having received the two products without knowing which he started with. A "wash-out" period of one week will be observed between the two administration periods to avoid so-called "carry-over" effects according to which the administration of the first drug could influence the effect of the second drug administered.
  Interventions: Drug: Ketamine 50 MG/ML; Drug: Esketamine 25 MG/ML
- BA group (Other): If A = Ketamine and B = Esketamine, each patient included in the study will be randomized in a sequence of administration of the two products. The BA sequence consists of patients starting with intravenous Esketamine 0,15 mg/kg in 1 hour (2 infusions separated by 6 weeks; Period 1) and continuing with intravenous Ketamine 0,3 mg/kg in 1 hour (2 infusions separated by 6 weeks; Period 2). Each patient will be monitored during the IV perfusion, and then, the next hour.
  The patient will receive a total of two infusions of Esketamine and then two infusions of Ketamine. Each patient will be his own witness because having received the two products without knowing which he started with. A "wash-out" period of one week will be observed between the two administration periods to avoid so-called "carry-over" effects according to which the administration of the first drug could influence the effect of the second drug administered.
  Interventions: Drug: Ketamine 50 MG/ML; Drug: Esketamine 25 MG/ML

INTERVENTIONS:
Drug: Ketamine 50 MG/ML — Intravenous Ketalar® 0,30 mg/kg in 1 hour.
Drug: Esketamine 25 MG/ML — Intravenous Vesierra® 0,15mg/kg in 1 hour.

SUMMARY:
Ketamine and Esketamine intravenous perfusions can modulate chronic pain. The purpose of this study is to determine if Ketamine or Esketamine are favorable for outpatients suffering from fibromyalgia.

DETAILED DESCRIPTION:
Ketamine and Esketamine intravenous perfusions in Pain Clinic can modulate chronic pain and are therefore part of the therapeutic arsenal of the Anesthesiologist in pain management. Patients with fibromyalgia syndrome have elevated levels of glutamate in the brain. This is demonstrated by functional brain imaging techniques. Elevation of glutamate is demonstrated in the posterior insular cortex, positively correlating with lower pain thresholds which is a hallmark of fibromyalgia syndrome. Ketamine has (e.a.) an inhibitory role of the N-methyl-D-aspartate (NMDA) receptor: it is a non-competitive antagonist of the NMDA receptor. In this context, Esketamine is available recently. This is the levorotatory form of Ketamine.

The main objective of this study is to measure if there is a difference between Ketamine and Esketamine on patients with fibromyalgia syndrome via the fibromyalgia impact questionnaire (FIQ) and measurement of side effects after intravenous perfusion. The fibromyalgia impact questionnaire is a global assessment of symptoms: pain, function, fatigue, stiffness, discomfort when walking up stairs, difficulties at work, anxiety, depression, days not worked and days of good quality in the past week.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Between 18 and 75 years old
* Reads and writes French
* Diagnosis of fibromyalgia syndrome according to Widespread Pain Index (WPI) and Symptom Severity Scale (SSS) score ≥ 13/31
* Both molecules (Ketamine and Esketamine) were administered at least once during an analgesic infusion session in Pain Clinic
* Patient with regular medical follow-up by a pain specialist at least 3 times a year

Exclusion Criteria:

* Allergy or intolerance to Ketamine or Esketamine
* Current infection, fever
* Pregnant or breastfeeding woman
* Serious cardiovascular disorders and severe hypertension
* Increased pressure of cerebrospinal fluid and severe intracranial disease
* Acute intermittent porphyria
* Untreated epilepsy
* Untreated glaucoma
* Difficult or impossible intravenous access
* Chronic Liver Disease Child-Pugh C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Score variations of Fibromyalgia Impact Questionnaire | At day 0 before starting each intravenous perfusion.
  Fibromyalgia Impact Questionnaire (FIQ) completed by the patient. The FIQ was developed from information gathered from patient reports, functional status instruments, and clinical observations. This instrument measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week. The score is between 0 and 100. In the severity analysis a FIQ total score from 0 to < 39 was found to represent a mild effect, ≥ 39 to < 59 a moderate effect, and ≥ 59 to 100 a severe effect.
Score variations of Fibromyalgia Impact Questionnaire | At day 7 after each intravenous perfusion.
  Fibromyalgia Impact Questionnaire (FIQ) completed by the patient. The FIQ was developed from information gathered from patient reports, functional status instruments, and clinical observations. This instrument measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week. The score is between 0 and 100. In the severity analysis a FIQ total score from 0 to < 39 was found to represent a mild effect, ≥ 39 to < 59 a moderate effect, and ≥ 59 to 100 a severe effect.
Score variations of Fibromyalgia Impact Questionnaire | At day 14 after each intravenous perfusion.
  Fibromyalgia Impact Questionnaire (FIQ) completed by the patient. The FIQ was developed from information gathered from patient reports, functional status instruments, and clinical observations. This instrument measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week. The score is between 0 and 100. In the severity analysis a FIQ total score from 0 to < 39 was found to represent a mild effect, ≥ 39 to < 59 a moderate effect, and ≥ 59 to 100 a severe effect.
Score variations of Fibromyalgia Impact Questionnaire | At day 21 after each intravenous perfusion.
  Fibromyalgia Impact Questionnaire (FIQ) completed by the patient. The FIQ was developed from information gathered from patient reports, functional status instruments, and clinical observations. This instrument measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week. The score is between 0 and 100. In the severity analysis a FIQ total score from 0 to < 39 was found to represent a mild effect, ≥ 39 to < 59 a moderate effect, and ≥ 59 to 100 a severe effect.
Score variations of Fibromyalgia Impact Questionnaire | At day 28 after each intravenous perfusion.
  Fibromyalgia Impact Questionnaire (FIQ) completed by the patient. The FIQ was developed from information gathered from patient reports, functional status instruments, and clinical observations. This instrument measures physical functioning, work status (missed days of work and job difficulty), depression, anxiety, morning tiredness, pain, stiffness, fatigue, and well-being over the past week. The score is between 0 and 100. In the severity analysis a FIQ total score from 0 to < 39 was found to represent a mild effect, ≥ 39 to < 59 a moderate effect, and ≥ 59 to 100 a severe effect.

SECONDARY OUTCOMES:
Heart rate disturbances after intravenous perfusion of Ketamine or Esketamine | At the beginning (minute zero) of each intravenous perfusion.
  Measurement of heart rate in Pain clinic during intravenous perfusion. Measurement in beat per minute.
Heart rate disturbances after intravenous perfusion of Ketamine or Esketamine | After 30 minutes of each intravenous perfusion.
  Measurement of heart rate in Pain clinic during intravenous perfusion. Measurement in beat per minute.
Heart rate disturbances after intravenous perfusion of Ketamine or Esketamine | After 60 minutes of each intravenous perfusion.
  Measurement of heart rate in Pain clinic during intravenous perfusion. Measurement in beat per minute.
Heart rate disturbances after intravenous perfusion of Ketamine or Esketamine | After 90 minutes of each intravenous perfusion.
  Measurement of heart rate in Pain clinic during intravenous perfusion. Measurement in beat per minute.
Heart rate disturbances after intravenous perfusion of Ketamine or Esketamine | After 120 minutes of each intravenous perfusion.
  Measurement of heart rate in Pain clinic during intravenous perfusion. Measurement in beat per minute.
Variations of Visual Analogue Scale for pain. | At the beginning (minute zero) of each intravenous perfusion.
  Measurement of Visual Analogue Scale (VAS) for pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Variations of Visual Analogue Scale for pain. | After 30 minutes of each intravenous perfusion.
  Measurement of Visual Analogue Scale (VAS) for pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Variations of Visual Analogue Scale for pain. | After 60 minutes of each intravenous perfusion.
  Measurement of Visual Analogue Scale (VAS) for pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Variations of Visual Analogue Scale for pain. | After 90 minutes of each intravenous perfusion.
  Measurement of Visual Analogue Scale (VAS) for pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Variations of Visual Analogue Scale for pain. | After 120 minutes of each intravenous perfusion.
  Measurement of Visual Analogue Scale (VAS) for pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Variations of Visual Analogue Scale for nausea. | At the beginning (minute zero) of each intravenous perfusion.
  Measurement of Visual Analogue Scale (VAS) for nausea. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no nausea" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater nausea.
Variations of Visual Analogue Scale for nausea. | After 30 minutes of each intravenous perfusion.
  Measurement of Visual Analogue Scale (VAS) for nausea. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no nausea" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater nausea.
Variations of Visual Analogue Scale for nausea. | After 60 minutes of each intravenous perfusion.
  Measurement of Visual Analogue Scale (VAS) for nausea. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no nausea" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater nausea.
Variations of Visual Analogue Scale for nausea. | After 90 minutes of each intravenous perfusion.
  Measurement of Visual Analogue Scale (VAS) for nausea. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no nausea" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater nausea.
Variations of Visual Analogue Scale for nausea. | After 120 minutes of each intravenous perfusion.
  Measurement of Visual Analogue Scale (VAS) for nausea. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no nausea" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater nausea.
Variations of non-invasive blood pressure. | At the beginning (minute zero) of each intravenous perfusion.
  Measurement of variations of systolic and diastolic non-invasive blood pressure with upper arm cuff. Measurement in mmHg.
Variations of non-invasive blood pressure. | After 30 minutes of each intravenous perfusion.
  Measurement of variations of systolic and diastolic non-invasive blood pressure with upper arm cuff. Measurement in mmHg.
Variations of non-invasive blood pressure. | After 60 minutes of each intravenous perfusion.
  Measurement of variations of systolic and diastolic non-invasive blood pressure with upper arm cuff. Measurement in mmHg.
Variations of non-invasive blood pressure. | After 90 minutes of each intravenous perfusion.
  Measurement of variations of systolic and diastolic non-invasive blood pressure with upper arm cuff. Measurement in mmHg.
Variations of non-invasive blood pressure. | After 120 minutes of each intravenous perfusion.
  Measurement of variations of systolic and diastolic non-invasive blood pressure with upper arm cuff. Measurement in mmHg.
Variations of pulse Oxygen saturation. | At the beginning (minute zero) of each intravenous perfusion.
  Measurement of variations of pulse Oxygen saturation (SpO2). Pulse oximetry is a non-invasive measures of oxygen saturation level in %. A normal SpO2 is typically between 95 and 100 percent. A SpO2 < 95 percent is considered low.
Variations of pulse Oxygen saturation. | After 30 minutes of each intravenous perfusion.
  Measurement of variations of pulse Oxygen saturation (SpO2). Pulse oximetry is a non-invasive measures of oxygen saturation level in %. A normal SpO2 is typically between 95 and 100 percent. A SpO2 < 95 percent is considered low.
Variations of pulse Oxygen saturation. | After 60 minutes of each intravenous perfusion.
  Measurement of variations of pulse Oxygen saturation (SpO2). Pulse oximetry is a non-invasive measures of oxygen saturation level in %. A normal SpO2 is typically between 95 and 100 percent. A SpO2 < 95 percent is considered low.
Variations of pulse Oxygen saturation. | After 90 minutes of each intravenous perfusion.
  Measurement of variations of pulse Oxygen saturation (SpO2). Pulse oximetry is a non-invasive measures of oxygen saturation level in %. A normal SpO2 is typically between 95 and 100 percent. A SpO2 < 95 percent is considered low.
Variations of pulse Oxygen saturation. | After 120 minutes of each intravenous perfusion.
  Measurement of variations of pulse Oxygen saturation (SpO2). Pulse oximetry is a non-invasive measures of oxygen saturation level in %. A normal SpO2 is typically between 95 and 100 percent. A SpO2 < 95 percent is considered low.

CONTACTS AND LOCATIONS:
Overall Officials: Brice Constant, MD, Principal Investigator — Centre Universitaire de Charleroi
Locations (1):
- CHU de Charleroi, Lodelinsart, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No
IPD will be available according to reasonable demands.